CLINICAL TRIAL: NCT05713422
Title: Superiority of Perineoplasty as Concomitant Surgical Procedure During Pelvic Organ Prolapse Repair; a Comparative Cohort Trial (SUPPORT)
Brief Title: Superiority of Perineoplasty as Concomitant Surgical Procedure During Pelvic Organ Prolapse Repair
Acronym: SUPPORT
Status: Active, not recruiting | Type: Observational
Sponsor: Marjolein Spiering (Other)
Collaborators: Spaarne Gasthuis (Other)
Responsible Party: Sponsor-Investigator, Marjolein Spiering, MSc, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL82381.018.22
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: POP; prolapse; perineoplasty
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative procedure; standard treatment: Vaginal level I and/or level II repair will be performed as usual (eg anterior and/or posterior colporrhaphy, sacrospinous fixation etc.) without perineoplasty as decided by surgeon and patient. This procedure is considered as the control group.
- Operative procedure; standard treatment including level III repair: Vaginal level I and/or level II repair will be performed as usual, but now including perineoplasty (level III repair) as decided by surgeon and patient. The decision of a perineoplasty to vaginal level I and/or level II repair is based on a shared decision made by surgeon together with the patient. The considerations upon which this decision has been established in a consensus meeting of Dutch urogynecologists and will be collected by a questionnaire, This group is considered as the 'intervention' group.

SUMMARY:
The goal of this study is to evaluate whether adding perineoplasty is, in comparison to performing vaginal prolapse surgery without adding perineoplasty, superior with respect to efficacy and cost-effectiveness and non-inferior with respect to morbidity, in patients undergoing vaginal surgical correction of pelvic organ prolapse at 24 months after surgery.

DETAILED DESCRIPTION:
Preoperative measurements, performed at baseline:

* Patient characteristics (age, BMI, smoking, obstetric history)
* Physical examination including POP-Q score. The genital hiatus (gh) at rest (as part of the POP-Q) will be used to assess the wideness of the vaginal introitus.
* Pelvic Floor Distress Inventory (PFDI-20) questionnaire and Patient Global Impression of Severity (PGI-S)
* Pelvic Floor Ultrasound 2DStudy measurements;
* Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-ir), Dutch Perineal Support Questionnaire (DPSQ), General Quality of Life (EQ-5D-5L), Medical Consumption Questionnaire (iMCQ) and Productivity Cost Questionnaire (iPCQ)
* Patient and surgeons considerations with respect to level III repair;

Postoperative measurements:

* Regular physical check-up will be at 4-8 weeks after procedure.
* Physical examination including POP-Q score
* Patient Global Impression of Improvement score (PGI-I)
* Pelvic Floor Ultrasound 2D
* iMCQ, iPCQ, EQ-5D-5L questionnaire

Extra follow up:

* Physical check-up 12 & 24 months after surgery:
* Physical examination including POP-Q score
* Pelvic Floor Ultrasound 2D
* PFDI-20, PGI-I, DPSQ, PISQ-ir, iMCQ, iPCQ, EQ-5D-5L questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Female patient >18 years of age
2. Complaints of pelvic organ prolapse
3. Indication for prolapse surgery (level I and/or level II repair)
4. Genital hiatus (GH) according to POP-Q staging of ≥4 cm and ≤7 cm

Exclusion Criteria:

1. Unable to understand the Dutch language
2. Pregnancy at baseline or intendancy to become pregnant during the study period
3. Patients with previous surgery for POP (previous mid urethral sling operations for urinary stress incontinence not excluded)
4. Unwilling and / or incapable of giving informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female organs
Study Population: Patients indicated for vaginal pelvic organ prolapse surgery.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Surgical success | 12 months
  composite outcome defined as meeting the 3 following conditions: [1] "much improved" or "improved" in response to the patient global impression of improvement questionnaire, [2] no re-intervention performed in the same compartment within the first 12 months after index surgery, [3] no stage 2 or more POP in the operated compartment.

SECONDARY OUTCOMES:
Morbidity | 24 months
  complications and re-interventions due to complications, pain
Effectiveness | 24 months
  disease specific and general quality of life
Anatomical outcomes | 24 months
Societal costs | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Spaarne Gasthuis, Haarlem
  - Bergman Clinics, Hilversum